CLINICAL TRIAL: NCT00003224
Title: Phase I Protocol for the Evaluation of the Safety and Immunogenicity of Vaccination With a Synthetic Melanoma Peptide in Patients With High Risk Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Craig L Slingluff, Jr, Professor of Surgery, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6346; NCI-H98-0010
Record Dates: First submitted 1999-11-01; First posted 2004-08-25 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — saponin QA-21V1; incomplete Freund's adjuvant; montanide ISA 51; peptide 946; gp100 Melanoma Antigen; gp100(280-288) melanoma antigen peptide; Tet-p peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: peptide 946 plus QS-21 (Experimental): 100 mcg peptide gp100 [280-288] plus 0.2 ml (100 mcg) QS-21 vaccine adjuvant
  Interventions: Biological: QS21; Biological: p946
- Group 2. p946 plus IFA (Experimental): 100 mcg peptide gp100 [280-288] plus 0.5 ml IFA (Montanide ISA-51) vaccine adjuvant
  Interventions: Biological: IFA (incomplete Freund's adjuvant); Biological: p946
- Group 3: p946 plus Tet-p plus QS-21 (Experimental): 100 mcg peptide gp100 [280-288],190 mcg tetanus peptide, plus 0.2 ml (100 mcg) QS-21 vaccine adjuvant
  Interventions: Biological: QS21; Biological: p946; Biological: Tet-p
- Group 4. p946, Tet-p plus IFA (Experimental): 100 mcg peptide gp100 [280-288], 190 mcg tetanus peptide, plus 0.5 ml IFA (Montanide ISA-51) vaccine adjuvant
  Interventions: Biological: IFA (incomplete Freund's adjuvant); Biological: p946; Biological: Tet-p
- Group 5: p946/Tet-p plus QS-21 (Experimental): 282 mcg gp100 [280-288]/tetanus peptide conjugate, plus 0.2 ml (100 mcg) QS-21 vaccine adjuvant
  Interventions: Biological: QS21; Biological: p946/tet-p
- Group 6. p946/Tet-p plus IFA (Experimental): 282 mcg gp100 [280-288]/tetanus peptide conjugate, plus 0.5 ml IFA (Montanide ISA-51) vaccine adjuvant
  Interventions: Biological: IFA (incomplete Freund's adjuvant); Biological: p946/tet-p

INTERVENTIONS:
Biological: QS21 — vaccine adjuvant
  Arms: Group 1: peptide 946 plus QS-21; Group 3: p946 plus Tet-p plus QS-21; Group 5: p946/Tet-p plus QS-21
Biological: IFA (incomplete Freund's adjuvant) — Peptides emulsified in IFA.
  Other Names: Montanide ISA-51, from Seppic.
  Arms: Group 2. p946 plus IFA; Group 4. p946, Tet-p plus IFA; Group 6. p946/Tet-p plus IFA
Biological: p946 — This a nonamer peptide YLEPGPVTA from Gp100, used as a melanoma vaccine antigen.
  Other Names: peptide 946, gp100 [280-288], YLEPGPVTA
  Arms: Group 1: peptide 946 plus QS-21; Group 2. p946 plus IFA; Group 3: p946 plus Tet-p plus QS-21; Group 4. p946, Tet-p plus IFA
Biological: p946/tet-p — This peptide is a longer version of p946 (gp100 [280-288]) sythesized colinearly with the tetanus helper peptide (Tet-p)
  Other Names: peptide 946-tetanus peptide conjugate melanoma vaccine
  Arms: Group 5: p946/Tet-p plus QS-21; Group 6. p946/Tet-p plus IFA
Biological: Tet-p — modified form of the p2 peptide from tetanus toxoid, used as nonspecific epitope for helper T cells.
  Other Names: tetanus peptide melanoma vaccine
  Arms: Group 3: p946 plus Tet-p plus QS-21; Group 4. p946, Tet-p plus IFA

SUMMARY:
RATIONALE: Vaccines made from peptide 946 may make the body build an immune response to kill tumor cells. Combining these vaccines with proteins from the tetanus vaccine, and/or with either QS21 or Montanide ISA-51 may be an effective treatment for metastatic melanoma.

PURPOSE: Randomized phase I trial to study the effectiveness of vaccines made from peptide 946 with or without tetanus peptide, QS21, or Montanide ISA-51 in treating patients with metastatic melanoma that cannot be surgically removed or with melanoma that is likely to recur.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the safety of peptide 946 melanoma vaccine (peptide 946), peptide 946 combined with tetanus peptide melanoma vaccine, or peptide 946-tetanus peptide conjugate in patients with high risk melanoma.

II. Determine the immunogenicity of peptide 946 melanoma vaccine (peptide 946), peptide 946 combined with tetanus peptide melanoma vaccine, or peptide 946-tetanus peptide conjugate in patients with high risk melanoma.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 6 treatment arms: Arm I: Patients receive peptide 946 melanoma vaccine (peptide 946) emulsified with QS21 subcutaneously (SQ). Arm II: Patients receive peptide 946 emulsified with Montanide ISA-51 (ISA-51) SQ. Arm III: Patients receive peptide 946 combined with tetanus peptide melanoma vaccine (tetanus peptide) emulsified with QS21 SQ. Arm IV: Patients receive peptide 946 combined with tetanus peptide emulsified with ISA-51 SQ. Arm V: Patients receive peptide 946-tetanus peptide conjugate emulsified with QS21 SQ. Arm VI: Patients receive peptide 946-tetanus peptide conjugate emulsified with ISA-51 SQ. Initially, 4 patients are randomized to Arm I and 4 patients are randomized to Arm II. If no dose limiting toxicities are observed in these patients, then additional patients are randomized to arms III-VI. Patients in each arm receive vaccine on day 0 and at months 1, 2, 3, 6, 9, and 12. Patients are followed at 6 and 12 months.

PROJECTED ACCRUAL: A maximum of 36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed unresectable metastatic melanoma (AJCC stage III or IV) OR resected melanoma with high risk of recurrence or mortality (stage IIB and above)
* Age: 18 to 79
* Performance status: ECOG 0-2
* Life expectancy: Greater than 12 months
* Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL
* Hepatic: AST and ALT no greater than 2.5 times upper limit of normal (ULN) Bilirubin no greater than 2.5 times ULN Alkaline phosphatase no greater than 2.5 times ULN
* Renal: Creatinine no greater than 1.5 times ULN

Exclusion criteria:

* patients currently receiving cytotoxic chemotherapy or who have received that therapy within the preceding 3 months
* known or suspected allergies to any component of the treatment vaccine
* unresectable tumor llikely to cause symptoms and for which therapy is anticipated within 3 months.
* receiving acute treatment for seriouis infection within 14 days.
* Patients with bulky disease, or with multiple brain metastases, but solitary brain metastases treated successfully with surgery or gamma knife may be eligible.
* Any of the following with 3 months:
* agentes with putative immunomodulating activity (except NSAIDs)
* allergy desensitizing injections
* other investigational agents
* interferons
* corticosteroids
* any growth factors
* prior melanoma vaccinations
* pregnancy or the possibility of becoming pregnant on study
* medical contraindication or potential problems in complying with the requirements of the protocol.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1996-02; Primary Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Study Chair — University of Virginia
Locations (1):
- Cancer Center, University of Virginia HSC, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Slingluff CL Jr, Yamshchikov G, Neese P, Galavotti H, Eastham S, Engelhard VH, Kittlesen D, Deacon D, Hibbitts S, Grosh WW, Petroni G, Cohen R, Wiernasz C, Patterson JW, Conway BP, Ross WG. Phase I trial of a melanoma vaccine with gp100(280-288) peptide and tetanus helper peptide in adjuvant: immunologic and clinical outcomes. Clin Cancer Res. 2001 Oct;7(10):3012-24. PMID 11595689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were enrolled at the University of Virginia
Pre-assignment Details: no enrolled patients were excluded.
Period: Overall Study
Arm/Group | Group 1: Peptide 946 Plus QS-21 | Group 2. p946 Plus IFA | Group 3: p946 Plus Tet-p Plus QS-21 | Group 4. p946, Tet-p Plus IFA | Group 5: p946/Tet-p Plus QS-21 | Group 6. p946/Tet-p Plus IFA
Started | 4 | 5 | 4 | 2 | 4 | 3
Completed | 4 | 5 | 4 | 2 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Peptide 946 Plus QS-21 | Group 2. p946 Plus IFA | Group 3: p946 Plus Tet-p Plus QS-21 | Group 4. p946, Tet-p Plus IFA | Group 5: p946/Tet-p Plus QS-21 | Group 6. p946/Tet-p Plus IFA | Total
Number analyzed (Participants) | 4 | 5 | 4 | 2 | 4 | 3 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 4 | 1 | 3 | 1 | 14
  >=65 years | 1 | 3 | 0 | 1 | 1 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (17.1) | 59.6 (18.6) | 44.3 (16.8) | 59.5 (17.7) | 51.8 (14.9) | 69.3 (7.5) | 55.6 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 2 | 2 | 10
  Male | 3 | 3 | 2 | 1 | 2 | 1 | 12
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 4 | 2 | 4 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Safety: Grade 3 Adverse Events
Description: Adverse events are monitored according to NCI/DCT Common Toxicity Criteria
Time Frame: Up to 24 months after last vaccine
Measure: Number; unit: participants
Groups:
- All QS-21: The toxicities are grouped for those receiving the vaccine adjuvant QS-21.
- All Montanide ISA-51: The toxicities are grouped for those receiving the vaccine adjuvant IFA (Montanide ISA-51).
Arm/Group | All QS-21 | All Montanide ISA-51
Number analyzed (Participants) | 12 | 10
participants | 1 | 0

2. Secondary Outcome: Immunogenicity of Each Vaccine Regimen
Description: T cell responses to the p946 (gp100 [280-288]) peptide. All enrolled patients were assayed for immune response to the gp100 peptide by ELIspot assay after 14 days in vitro sensitization. The number with a response in each study arm is reported.
Time Frame: up to 12 months since enrollment
Measure: Number; unit: participants
Arm/Group | Group 1: Peptide 946 Plus QS-21 | Group 2. p946 Plus IFA | Group 3: p946 Plus Tet-p Plus QS-21 | Group 4. p946, Tet-p Plus IFA | Group 5: p946/Tet-p Plus QS-21 | Group 6. p946/Tet-p Plus IFA
Number analyzed (Participants) | 4 | 5 | 4 | 2 | 4 | 3
participants | 1 | 1 | 0 | 1 | 0 | 0

3. Other Pre Specified Outcome: Number of Participants With a Proliferative Response to Tetanus Helper Peptide
Description: Proliferative response measured in participants using a tritiated thymidine incorporation assay with peripheral blood mononuclear cells (PBMC) stimulated with the tetanus peptide in vitro, and measured at 5 days after in vitro culture.
Time Frame: during vaccination
Population: All evaluable enrolled patients were assayed.
Measure: Number; unit: participants
Arm/Group | Group 1: Peptide 946 Plus QS-21 | Group 2. p946 Plus IFA | Group 3: p946 Plus Tet-p Plus QS-21 | Group 4. p946, Tet-p Plus IFA | Group 5: p946/Tet-p Plus QS-21 | Group 6. p946/Tet-p Plus IFA
Number analyzed (Participants) | 3 | 5 | 3 | 2 | 4 | 3
participants | 1 | 0 | 1 | 2 | 4 | 2

ADVERSE EVENTS:
Description: Participants are reported for adverse events based on vaccine adjuvant received because the adverse events were considered primarily related to the adjuvant. Also, the gp100 peptide was included in all 6 study groups.
Groups:
- QS-21 Adjuvant: The combination of participants from Arms 1, 3, and 5, all treated with peptides plus QS-21 adjuvant
- Montanide ISA-51 Adjuvant: The combination of participants from Arms 2, 4, and 6, all treated with peptides plus Montanide ISA-51 adjuvant
Arm/Group | QS-21 Adjuvant | Montanide ISA-51 Adjuvant
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/10
Other Adverse Events (participants affected / at risk) | 11/12 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QS-21 Adjuvant (N=12) | Montanide ISA-51 Adjuvant (N=10)
Esophageal spasm, Grade 3 (Gastrointestinal disorders) | 1 | 0 — This occurred in one patient on group 3, whose vaccine incorporated QS-21.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QS-21 Adjuvant (N=12) | Montanide ISA-51 Adjuvant (N=10)
grade 1-2 skin toxicity, especially pain (Skin and subcutaneous tissue disorders) | 9 | 3 — vaccine site, typically transient.
skin, other (Skin and subcutaneous tissue disorders) | 4 | 0
Flu-like symptoms (General disorders) | 2 | 3
Headache (Nervous system disorders) | 3 | 1
Other pain (General disorders) | 2 | 0
other gastrointestinal (Gastrointestinal disorders) | 2 | 1
other neurological (Nervous system disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Hematological (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
endocrine (Endocrine disorders) | 0 | 1
Urinary (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes